CLINICAL TRIAL: NCT04121156
Title: The Effect of High Definition Transcranial Direct Current Stimulation (HD-tDCS) on Cognitive Function in Patients With Mild Cognitive Impairment: a Randomized, Triple-blind, Sham-controlled, Pilot Study
Brief Title: High Definition Transcranial Direct Current Stimulation (HD-tDCS) in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Che-Sheng Chu, Attending physician of department of psychiatry, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGHKS-2068
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 milli Amp dose of HD-tDCS treatment (Active Comparator): 2 milli Amp dose of HD-tDCS treatment for for 25 minutes, once working day for 2 weeks, total 10 sessions
  Interventions: Device: HD-tDCS treatment
- Sham (placebo) dose of HD-tDCS treatment (Sham Comparator): Sham (placebo) dose of HD-tDCS treatment for 25 minutes, once working day for 2 weeks, total 10 sessions
  Interventions: Device: sham (placebo) HD-tDCS

INTERVENTIONS:
Device: HD-tDCS treatment — 2 milli Amp dose of HD-tDCS treatment for for 20 minutes, for 5 consecutive twice daily sessions
  Arms: 2 milli Amp dose of HD-tDCS treatment
Device: sham (placebo) HD-tDCS — Participants will receive sham (placebo) HD-tDCS for 20 minutes, for 5 consecutive twice daily sessions
  Arms: Sham (placebo) dose of HD-tDCS treatment

SUMMARY:
The study aimed to investigate whether high definition transcranial direct current stimulation (HD-tDCS) could benefit global cognitive function and sub-domains of cognition (visual/verbal/working memory, executive function, attention, processing speed, language, and frontal lobe function), mood (depression and anxiety), and subjective memory impairment in patients with mild cognitive impairment.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS), a novel, non-invasive and safe neuro-modulating technique, has been developed as a new therapeutic option for neuropsychiatric disorders. It encompasses the induction of a relatively weak constant current flow through the cerebral cortex via scalp electrodes. Dependent on stimulation polarity, this results in a modulation of cortical excitability and spontaneous neural activity. Compared with tDCS, high-definition transcranial direct current stimulation (HD-tDCS) is highly focal and can specifically modulate cortical activity within the region confined by its 4 x 1 ring of elctrodes, such that the targeted region becomes more amenable to neuroplastic change. Studies have suggested that tDCS improve cognition, including memory recall, verbal fluency and executive function. Yet, there is not HD-tDCS study on MCI. The purpose of this study is to examine whether HD-tDCS could benefit global cognitive function and sub-domains of cognition (visual/verbal/working memory, executive function, attention, processing speed, language, and frontal lobe function), mood (depression and anxiety), and subjective memory impairment in patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 to 85 years
* mild cognitive impairment
* right handed

Exclusion Criteria:

* Having epilepsy, severe physical illness, any current psychiatric comorbidity or history of substance dependence
* Having contraindications for transcranial electrical/magnetic stimulation.
* Having intracranial metal foreign bodies
* Having a history of intracranial neoplasms or surgery, or a history of severe head injuries or cerebrovascular diseases
* Receiving psychotropic agents such as antipsychotic, antidepressant, benzodiazepam and anxiolytics etc.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Cognitive Abilities Screening Instrument, CASI | Change from baseline after one week, one and three months
  The Cognitive Abilities Screening Instrument (CASI) is a cognitive test screening for dementia, in monitoring the disease progression, and in providing profiles of cognitive impairment by examining abilities on attention, concentration, orientation, short-term memory, long-term memory, language abilities, visual construction, list-generating fluency, abstraction, and judgment with score ranges of 0 to 100, respectively.
Wechsler Memory Scale-third edition (WMS III) - verbal paired associates I and II | Change from baseline after one week, one and three months
  For assessing verbal memory by assessing recall memory for orally presented word pairs that have been previously learned (verbal paired associates I); assessing ability to recall associations from Verbal Paired Associates I after a 30-minute delay, as well as assessing recognition of word pairs (verbal paired associates II).
Wechsler Memory Scale-third edition (WMS III) - visual reproduction I and II | Change from baseline after one week, one and three months
  For assessing visual memory function by assessing ability to reproduce difficult-to-verbalize designs after a brief exposure (visual reproduction I); assessing ability to recall the designs presented in Visual Reproduction I after a 30-minute delay, as well as specific sub-subtests to assess recognition of correct figures from nontarget figures, copying of figures to assess visual perception abilities, and a subtest to analyze discrimination abilities (visual reproduction II).
Wisconsin card sorting test | Change from baseline after one week, one and three months
  for assessing executive function
Frontal assessment battery, FAB | Change from baseline after one week, one and three months
  The FAB is a brief tool that can be used at the bedside or in a clinic setting to assist frontal function of subjects. Total score is from a maximum of 18, higher scores indicating better performance. The scales consist similarities (conceptualization), lexical fluency (mental flexibility), motor series "Luria" test (programming), conflicting instructions (sensitivity to interference), Go-No Go (inhibitory control), prehension behaviour (environmental autonomy).
Wechsler adult intelligence scale four edition, WAIS-IV, digit span | Change from baseline after one week, one and three months
  The Wechsler Adult Intelligence Scale (WAIS) is an IQ test designed to measure intelligence and cognitive ability in adults and older adolescents. It is currently in its fourth edition (WAIS-IV) released in 2008 by Pearson, and is the most widely used IQ test, for both adults and older adolescents, in the world.
  We used WAIS-IV, digit span subscale, to examine attention among subjects; Digit span was by listening to sequences of numbers orally and to repeat them as heard, in reverse order, and in ascending order.
Wechsler adult intelligence scale four edition, WAIS-IV, digit symbol coding | Change from baseline after one week, one and three months
  We used WAIS-IV, digit symbol coding subscale, to examine processing speed among subjects; The digit symbol coding is a paper-and-pencil cognitive test presented on a single sheet of paper that requires a subject to match symbols to numbers according to a key located on the top of the page. The subject copies the symbol into spaces below a row of numbers. The number of correct symbols within the allowed time, usually 90 to 120 seconds, constitutes the score
Wechsler adult intelligence scale four edition, WAIS-IV, vocabulary | Change from baseline after one week, one and three months
  We used WAIS-IV, vocabulary subscale, to examine language function among subjects; The vocabulary subtest requires the client to try to define up to 30 words. This subtest assesses the client's understanding of words and reflects: language development, expressive language skills, cultural and educational experiences, ability to use words appropriately, retrieval of information from long-term memory.

SECONDARY OUTCOMES:
Beck depression inventory (BDI-II) | Change from baseline after one week, one and three months
  The BDI-II was a 1996 revision of the BDI. Participants were asked to rate how they have been feeling for the past two weeks. BDI-II also contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Beck anxiety inventory (BAI) | Change from baseline after one week, one and three months
  The Beck Anxiety Inventory (BAI), created by Aaron T. Beck and other colleagues, is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are as follows: 0-7: minimal anxiety; 8-15: mild anxiety; 16-25: moderate anxiety; 26-63: severe anxiety.
Subjective Cognitive Decline Questionnaire (SCD-Q MyCog) | Change from baseline after one week, one and three months
  The SCD-Q is a validated questionnaire that assesses the presence of a subjective cognitive decay in abilities such as memory, attention, language or executive functions. This scale is made up of two parts: MyCog is filled by the subject, TheirCog by the caregiver. Both parts have 24 identical dichotomous questions (yes/no), that evaluate decline for memory performances, language and executive functions in the last 2 years of daily life. The SCD-Q score for MyCog and TheirCog ranges from 0 to 24, with higher scores associated with greater perceived cognitive changes (cut to be classified as SCD = 7).

CONTACTS AND LOCATIONS:
Overall Officials: Che-Sheng Chu, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Department of Psychiatry, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chu CS, Chang HA, Lin YT, Shen HC, Liang CK, Hsu YH, Pan CC, Kuo HY, Liang WZ, Chen SL, Chen CS. Effectiveness and safety of high-definition transcranial direct current stimulation in patients with mild cognitive impairment: A randomized, triple-blind, sham-controlled trial. J Alzheimers Dis. 2025 Nov;108(1):298-311. doi: 10.1177/13872877251376547. Epub 2025 Sep 22. PMID 40984052